CLINICAL TRIAL: NCT00402844
Title: A Multicenter Clinical Safety Assessment of Polypropylene Transvaginal Mesh in Pelvic Reconstructive Surgery
Brief Title: Safety Study of Pelvic Organ Prolapse Repair Using Transvaginal Mesh
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TVM-II-2006
Record Dates: First submitted 2006-11-20; First posted 2006-11-22 (Estimated); Last update posted 2007-11-14 (Estimated); Status verified 2007-11

CONDITIONS: Pelvic Organ Prolapse
Keywords: Multicenter; Pelvic organ prolapse; Prospective; Transvaginal mesh
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Transvaginal mesh- PROLIFT®-system

SUMMARY:
Pelvic organ prolapse is characterized by a lack of pelvic floor support causing the pelvic organs and vaginal walls to protrude. For decades, suture repair techniques have been the primary choice of surgical treatment when indicated.

The notion of reinforcing pelvic floor defects using biomaterial implants is not an exclusively contemporary idea. Traditional surgical techniques are frequently associated with unsatisfying anatomical recurrence rates and over the years sporadic attempts have been made to introduce novel surgical techniques using a variety of biomaterials as support with varying success. It is plausible that inherently weak, or damaged, pelvic floor supportive tissues need to be reinforced by a permanent support to avoid the high rates of recurrences commonly described using traditional techniques. However, use of biomaterials in pelvic reconstructive surgery has become widespread in just a few years despite a lack of clinical safety data, or compelling clinical evidence demonstrating that it improves outcomes compared to traditional suture techniques.

It is likely that biomaterials need to be "anchored" in tissues not afflicted by the disease, in order to provide the intended pelvic floor support. This has given rise to transvaginal surgical techniques using a transobturator approach passing the mesh through the arcus tendineous fascia pelvis, or the sacrospinous ligaments through a transgluteal approach. Already commercially available implant materials are in need of patient safety documentation, both when considering the surgical techniques by which these materials are placed in the body as well as the actual materials. Complication rates and perioperative morbidity using these surgical routes in pelvic organ prolapse surgery are generally unknown.

The aim of the present study was to assess the long term morbidity, and describe the complications, associated with transvaginal mesh repair of pelvic organ prolapse using the PROLIFT®-system.

DETAILED DESCRIPTION:
Main objective:

- To describe short and long-term complications associated with pelvic organ prolapse repair using macroporous polypropylene transvaginal mesh (TVM) using a transobturator or transgluteal approach.

Secondary objectives:

* To describe anatomical restoration of the pelvic floor following transvaginal mesh repair of pelvic organ prolapse using the Pelvic Organ Prolapse Quantification system (POP-Q).
* To describe subjective patient outcomes using validated questionnaires with regard to pelvic organ function (UDI), sexual function (PISQ) and quality of life (IIQ).

Study design:

- A prospective multicenter open labeled single cohort study.

Study protocol:

* At baseline patients receive oral and written information about the study.
* Following informed consent, patients are included in the study if pelvic organ prolapse surgery is indicated and all inclusion, and no exclusion, criteria are fulfilled.
* Preoperatively all patients answer a detailed self reported questionnaire on health history, previous surgery, obstetrical history and current diseases and medications. The questionnaire also includes questions on symptoms from the pelvic organs and pelvic floor.
* Preoperatively all patients undergo a clinical examination using the POP-Q system, as well as, a validated clinical inflammatory grading of the vaginal compartments.
* Patients undergo the TVM procedure in a standardised manner with all participating surgeons having undergone pretrial surgical training and adopting the same surgical technique. All patients receive standardised intraoperative antibiotics.
* Complications during the immediate peri- and postoperative hospital stay are registered in hospital charts.
* All patients receive a clinical follow-up appointment 2 months, 1 year and 3 years after surgery. At follow-up identical self reported questionnaires are used for subjective assessment. Clinical examinations are performed as preoperatively suing the POP-Q system and macroscopic inflammatory grading. Complications are registered in a specific protocol and hospital charts.
* All protocols are to be submitted after the 2 months follow-up for an interrim safety analysis. The study chair is responsible for stopping the study if the rate, or seriousness, of complications exceed the expected.
* Patients are free to withdraw from the study at any point.

ELIGIBILITY:
Inclusion Criteria:

* Pelvic organ prolapse stage 2 or more according to the POP-Q staging system
* Symptoms related to pelvic organ prolapse including bulging, pelvic heaviness and vaginal protrusion
* Able to make an informed consent to participate
* Physically and mentally able to participate in follow-up

Exclusion Criteria:

* Previous pelvic organ cancer regardless of treatment
* Severe rheumatic disease requiring per oral steroid treatment
* Systemic connective tissue disorder (SLE, Sjögrens syndrome, Marfans syndrome, Ehlers Danhlos, collagenosis, polymyositis or polymyalgia rheumatica)
* Physically or mentally unable to participate in follow-up or give informed consent to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250
Dates: Start 2006-08; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Immediate and delayed TVM-related complications. | 1 year

SECONDARY OUTCOMES:
Anatomical outcome using the validated POP-Q staging system. | 1 year
Subjective outcome using the validated UDI, IIQ and PISQ. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Altman, MD, PhD, Study Chair — Karolinska Institutet
Locations (26):
- Denmark (2):
  - Nyköbing Hospital, Nyköbing
  - Skejby Hospital, Skejby
- Finland (4):
  - Jorvi Hospital, Jorvi
  - Lahti Hospital, Lahti
  - Lojo Hospital, Lohja
  - Åbo Hospital, Turku
- Norway (7):
  - Akershus University Hospital, Ahus
  - Haukeland Hospital, Bergen
  - Bærum Hospital, Bærum
  - Gjøvik Hospital, Gjøvik
  - Kongsberg Hospital, Kongsberg
  - Rikshospitalet, Oslo
  - The Regional Hospital in Tromsø, Tromsø
- Sweden (13):
  - Sahlgrenska Hospital, Gothenburg
  - Halmstad Hospital, Halmstad
  - Kristiansstad Hospital, Kristiansstad
  - Linköping University Hospital, Linköping
  - Vrinnevi Hospital, Norrköping
  - Örebro University Hospital, Örebro
  - Skaraborg Hospital Skövde, Skövde
  - Danderyd University Hospital, Stockholm
  - S:t Göran Hospital, Stockholm
  - South Hospital, Stockholm
  - Uppsala Academic Hospital, Uppsala
  - Västerås Hospital, Västerås
  - Ystad Hospital, Ystad

REFERENCES:
- [Background] Altman D, Falconer C. Perioperative morbidity using transvaginal mesh in pelvic organ prolapse repair. Obstet Gynecol. 2007 Feb;109(2 Pt 1):303-8. doi: 10.1097/01.AOG.0000250970.23128.63. PMID 17267828
- [Derived] Elmer C, Falconer C, Hallin A, Larsson G, Ek M, Altman D; Nordic Transvaginal Mesh Group. Risk factors for mesh complications after trocar guided transvaginal mesh kit repair of anterior vaginal wall prolapse. Neurourol Urodyn. 2012 Sep;31(7):1165-9. doi: 10.1002/nau.22231. Epub 2012 Apr 19. PMID 22517125
- [Derived] Altman D, Elmer C, Kiilholma P, Kinne I, Tegerstedt G, Falconer C; Nordic Transvaginal Mesh Group. Sexual dysfunction after trocar-guided transvaginal mesh repair of pelvic organ prolapse. Obstet Gynecol. 2009 Jan;113(1):127-133. doi: 10.1097/AOG.0b013e3181922362. PMID 19104368
- [Derived] Elmer C, Altman D, Engh ME, Axelsen S, Vayrynen T, Falconer C; Nordic Transvaginal Mesh Group. Trocar-guided transvaginal mesh repair of pelvic organ prolapse. Obstet Gynecol. 2009 Jan;113(1):117-126. doi: 10.1097/AOG.0b013e3181922164. PMID 19104367
- [Derived] Altman D, Vayrynen T, Engh ME, Axelsen S, Falconer C; Nordic Transvaginal Mesh Group. Short-term outcome after transvaginal mesh repair of pelvic organ prolapse. Int Urogynecol J Pelvic Floor Dysfunct. 2008 Jun;19(6):787-93. doi: 10.1007/s00192-007-0526-2. PMID 18074068